CLINICAL TRIAL: NCT00130364
Title: Efficacy and Safety of Pimecrolimus Cream 1% in Patients (2 to 11 Years Old) With Mild to Moderate Facial Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981C2440
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; T-cell; pimecrolimus; children; facial; Facial atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Facies | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Pimecrolimus vehicle cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus 1 % cream
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Pimecrolimus vehicle cream (placebo)
  Arms: 2

SUMMARY:
This study is not being conducted in the United States of America (USA).

Atopic dermatitis, also called eczema, is characterized by redness, papulation (skin elevation) and pruritus (skin itching). The active ingredient of pimecrolimus inhibits T-cell activation. These cells are involved in the inflammatory component of the disease. This study will test the safety and efficacy of pimecrolimus cream 1% in atopic dermatitis of the face in patients intolerant of, or dependent on, topical corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate facial atopic dermatitis
* Patients intolerant of, or dependent on, topical corticosteroids

Exclusion Criteria:

* Concurrent skin diseases (infections)
* Immunocompromised
* Recently received phototherapy or systemic therapy

Ages: 2 Years to 11 Years | Sex: All
Age Groups: Child
Enrollment: 200
Dates: Start 2005-08; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who have a facial Investigator's Global Assessment (IGA) score of 0 or 1 (clear or almost clear)

SECONDARY OUTCOMES:
Percentage of patients who responded to treatment assessed by overall Eczema Area and Severity Index (EASI) and head and neck EASI score
The percentage of patients achieving at least a 60 % reduction from baseline in the head and neck EASI score
The percentage of patients achieving a score of 0 or 1 for pruritus (absent or mild)
Time to clearance of facial IGA (score of 0 or 1)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- This study is not being conducted in the United States, Novartis Pharmaceuticals, New Jersey, United States